CLINICAL TRIAL: NCT00576303
Title: A Single-arm, Open Label Multicenter Study to Assess the Efficacy, Safety and Tolerability of Once Monthly Administration of C.E.R.A. for the Maintenance of Hemoglobin Levels in Dialysis Patients With Chronic Renal Anemia
Brief Title: A Study of Intravenous Mircera in Dialysis Patients With Chronic Renal Disease and Anemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20977
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- RO0503821 (C.E.R.A.), 1x/4weeks (Experimental): Eligible participants started RO0503821 (Continuous Erythropoietin Receptor Activator [C.E.R.A]) intravenously, at a dose of 120, 200 or 360 microgram (µg) every four weeks. The dose of C.E.R.A was based on the epoetin alfa or beta dose of<8000, 8000-16000, or >16000 international units (IU)/week, administered during the stability verification period (SVP) of 4 weeks. The SVP period was followed by dose titration period (DTP) of 16 weeks, efficacy evaluation period (EEP) of 8 weeks and long term safety period (LTSP) of 28 weeks
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120, 200 or 360 micrograms iv monthly (starting dose)

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of monthly intravenous Mircera for the maintenance of hemoglobin levels in dialysis patients with chronic renal disease, currently receiving epoetin alfa or beta. Patients will receive monthly intravenous injections of Mircera at a starting dose of 120, 200 or 360 micrograms/month, depending on the dose of epoetin alfa or beta they were receiving in the week preceding study start. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* hemodialysis or peritoneal dialysis, with same mode of dialysis for >=3 months before and throughout screening period;
* continuous maintenance epoetin alfa or beta therapy with the same dosing interval during the previous 2 months.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension requiring interruption of epoetin alfa or beta treatment in past 6 months;
* significant acute or chronic bleeding such as overt gastrointestinal bleeding;
* hemolysis;
* folic acid and vitamin B12 deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Russia (8):
  - Kemerovo
  - Krasnodar
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Volzhsky
  - Yekaterinburg

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 241 participants were recruited across 19 centers in Russia. The study was conducted from 29 Apr 2008 to 09 Jun 2010.
Pre-assignment Details: Of the 241 screened participants, 200 participants received the study drug and 41 participants were early withdrawals during the stability verification period (SVP)
Groups:
- RO0503821 (1x/4 Weeks): Eligible participants started RO0503821 (Continuous Erythropoietin Receptor Activator [C.E.R.A]) intravenously, at a dose of 120, 200 or 360 microgram (µg) every four weeks. The dose of C.E.R.A was based on the erythropoiesis stimulating agents (ESA) like epoetin alfa or beta dose of<8000, 8000-16000, or >16000 international units (IU)/week, administered during the stability verification period (SVP) of 4 weeks. The SVP period was followed by dose titration period (DTP) of 16 weeks, efficacy evaluation period (EEP) of 8 weeks and long term safety period (LTSP) of 28 weeks
Period: Dose Titration Period
Arm/Group | RO0503821 (1x/4 Weeks)
Started | 200
Completed | 183
Not Completed | 17
Not completed — Early withdrawal | 17
Period: Efficacy Evaluation Period
Arm/Group | RO0503821 (1x/4 Weeks)
Started | 183
Completed | 178
Not Completed | 5
Not completed — Early withdrawal | 5
Period: Long Term Safety Period
Arm/Group | RO0503821 (1x/4 Weeks)
Started | 178
Completed | 162
Not Completed | 16
Not completed — Early withdrawal | 16

BASELINE CHARACTERISTICS:
Groups:
- RO0503821 (1x/4 Weeks): Eligible participants started RO0503821 (C.E.R.A) intravenously, at a dose of 120, 200 or 360 µg every four weeks. The dose of C.E.R.A was based on the ESA like epoetin alfa or beta dose of <8000, 8000-16000, or >16000 IU/week, administered during the SVP of 4 weeks. The SVP was followed by DTP of 16 weeks, EEP of 8 weeks and LTSP of 28 weeks
Arm/Group | RO0503821 (1x/4 Weeks)
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Average Hemoglobin Concentration Within +- 1 Gram/Deciliter of Their Reference Hb and Between 10.5 and 12.5 Gram/Deciliter During EEP
Description: All mean Hb values recorded during the evaluation period were calculated and subtracted from the mean baseline Hb value for each participant. The percentage of participants maintaining their mean Hemoglobin (Hb) concentration within +/- 1 gram/deciliter (g/dL) of their reference Hb and between 10.5 -12.5 g/dL is presented during the EEP. The EEP is defined as Week 16 to Week 24
Time Frame: EEP (Week 16 to Week 24)
Population: Per protocol (PP) population included participants except who didn't meet inclusion criterion relative to consent, stable baseline Hb values, iron status, epoetin maintenance, and who met exclusion criterion of hemoglobinopathies/hemolysis, bleeding, >3 recorded Hb, missing drug administration, other ESA, blood transfusion during the DTP or EEP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RO0503821 (1x/4 Weeks)
Number analyzed (Participants) | 145
percentage of participants | 54.5 [46.0 to 62.8]

2. Secondary Outcome: Mean Change in Hb Concentration From Baseline to the EEP
Description: A time adjusted mean change in Hb concentration was calculated using an area under the curve approach, for both periods separately. Change in Hb concentration between the baseline and evaluation periods was calculated by subtracting the calculated average baseline Hb value from the average evaluation period Hb value. All blood samples for Hb measurements were taken prior to study drug administration. Analysis used last observation carried forward (LOCF) for missing Hb values to correct for the impact of early dropouts. The baseline period is defined as Week -4 to Week -1. The EEP is defined as Week 16 to Week 24
Time Frame: Baseline (Week -4 to Week -1), EEP (Week 16 to Week 24)
Population: The Intent-to-Treat (ITT) population included all the participants who received at least one dose of C.E.R.A. and for whom data for at least one follow-up variable is available.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | RO0503821 (1x/4 Weeks)
Number analyzed (Participants) | 199
g/dL | 0.19 (1.21)

3. Secondary Outcome: Percentage of Participants Maintaining Average Hb Concentration Within Target Range of 10.5-12.5 g/dL Throughout the EEP
Description: All mean Hb values recorded during the EEP were calculated. The percentage of participants maintaining their average Hb concentration within the targeted range 10.5-12.5 g/dL during the EEP were reported. The EEP is defined as Week 16 to Week 24
Time Frame: EEP (Week 16 to Week 24)
Population: The ITT population included all the participants who received at least one dose of C.E.R.A. and for whom data for at least one follow-up variable is available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RO0503821 (1x/4 Weeks)
Number analyzed (Participants) | 199
percentage of participants | 63.8 [56.7 to 70.5]

4. Secondary Outcome: Mean Number of Days Spent Within Hb Range of 10.5-12.5 g/dL During the EEP
Description: The mean number of days the participant spent within the Hb range 10.5-12.5 g/dL during the EEP was reported. The EEP is defined as Week 16 to Week 24
Time Frame: EEP (Week 16 to Week 24)
Population: The ITT population included all the participants who received at least one dose of C.E.R.A. and for whom data for at least one follow-up variable is available. Of the 199 participants, analysis was conducted on 184 participants, as 15 participants did not maintain their hemoglobin, within range of 10.5-12.5 g/dL during the EEP.
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | RO0503821 (1x/4 Weeks)
Number analyzed (Participants) | 184
number of days | 34.7 (18.42)

5. Secondary Outcome: Number of Participants Requiring Any Dose Adjustment During the DTP, EEP, and LTSP
Description: The number of participants who required dose adjustments of C.E.R.A were categorized as; 1. No dose change; 2. Any dose change: a. Dose increase only; b. Dose decrease only; c. Dose increase and increase; 3. Only one dose, all of which were recorded during DTP, EEP and LTSP. DTP is defined as Week 1 to Week 16, EEP is defined as Week 16 to Week 24 and LTSP is defined as Week 24 to Week 44
Time Frame: DTP (Week 1 to Week 16), EEP (Week 16 to Week 24) and LTSP (Week 24 to Week 44)
Population: The ITT population included all the participants who received at least one dose of C.E.R.A. and for whom data for at least one follow-up variable is available. . Data for the participants present at the time of assessment was used for analysis i.e. for DTP- 199, EEP-183, LTSP-178 respectively.
Measure: Number; unit: number of participants
Arm/Group | RO0503821 (1x/4 Weeks)
Number analyzed (Participants) | 199
number of participants
  DTP, No dose change | 50
  DTP, Dose increase only | 37
  DTP, Dose decrease only | 68
  DTP, Dose decrease and increase | 41
  DTP, Only one dose | 3
  EEP, No dose change | 81
  EEP, Dose increase only | 46
  EEP, Dose decrease only | 42
  EEP, Dose decrease and increase | 12
  EEP, Only one dose | 2
  LTSP, No dose change | 39
  LTSP, Dose increase only | 41
  LTSP, Dose decrease only | 55
  LTSP, Dose decrease and increase | 40
  LTSP, Only one dose | 3

6. Secondary Outcome: Number of Participants With Red Blood Cell Transfusion
Description: The number of participants who underwent red blood cell transfusion was reported
Time Frame: Up to 3 years
Population: The safety population was defined as all participants who received at least one dose of the trial medication and underwent a safety follow-up, whether withdrawn prematurely or not.
Measure: Number; unit: number of participants
Arm/Group | RO0503821 (1x/4 Weeks)
Number analyzed (Participants) | 200
number of participants | 5

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Serious adverse events and non-serious adverse events are reported in the safety population.
Arm/Group | RO0503821 (1x/4 Weeks)
Serious Adverse Events (participants affected / at risk) | 45/200
Other Adverse Events (participants affected / at risk) | 78/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/4 Weeks) (N=200)
Anaemia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 4
Death (General disorders) | 1
Device dislocation (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 3
Cholestasis (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Ear infection (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis chronic (Infections and infestations) | 1
Pyonephrosis (Infections and infestations) | 1
Renal cyst infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 14
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetic coma (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/4 Weeks) (N=200)
Anaemia (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Myopia (Eye disorders) | 1
Retinopathy hypertensive (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 5
Gastritis atrophic (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 4
Gastroduodenitis (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 2
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 4
Hiatus hernia (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 3
Periodontitis (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Chest pain (General disorders) | 1
Hyperthermia (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Pyelonephritis chronic (Infections and infestations) | 1
Pyonephrosis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Viral hepatitis carrier (Infections and infestations) | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Poisoning (Injury, poisoning and procedural complications) | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 2
Scapula fracture (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 2
Haemoglobin decreased (Investigations) | 1
Fluid retention (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Polydipsia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Hypotonia (Nervous system disorders) | 2
Intercostal neuralgia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Radiculitis cervical (Nervous system disorders) | 1
Radiculitis lumbosacral (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 2
Renal cyst (Renal and urinary disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 1
Aortic arteriosclerosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 16
Ischaemia (Vascular disorders) | 1
Post thrombotic syndrome (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.